CLINICAL TRIAL: NCT03789266
Title: Drains Ablation Post Total Hip Arthroplasty : Search for the Least Painful Technique
Acronym: TADDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2016/0382/HP
Record Dates: First submitted 2018-07-24; First posted 2018-12-28 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Total Hip Arthroplasty; Drain Insertion Site

STUDY DESIGN:
Who Masked: Participant
Masking Description: patient will not know which technique will be used for drain ablation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drain ablation - Non Aspiration mode (Experimental): Drain ablation will be done in non Aspiration mode
  Interventions: Procedure: drain ablation
- Drain ablation - Aspiration mode (Other): Drain ablation will be done in Aspiration mode
  Interventions: Procedure: drain ablation

INTERVENTIONS:
Procedure: drain ablation — drain ablation will be done in Aspiration mode or in non Aspiration mode

SUMMARY:
Comparison of ablation technique of drains

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted to the orthopedic surgery department for surgery for a total hip arthroplasty
2. Signed inform consent form

Exclusion Criteria:

1. Drain in non-aspirating mode at the time of medical ablation prescription
2. Administration of analgesic III in the 12 hours preceding the inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-03-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the pain felt by the patients at the time of the removal of the drain, using the pain visual analogue scale | 20 minutes
  pain will be measured using a visual analogic scale from 0 (for no pain) to 10 (fo maximum pain)

SECONDARY OUTCOMES:
Presence of haematoma after ablation | Day 2 post ablation
  Presence or absence of haematoma will be visually checked

CONTACTS AND LOCATIONS:
Overall Officials: Mylène BONNAIRE, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No